CLINICAL TRIAL: NCT00925613
Title: Exchange of a Double Lumen Tube With a Proseal Laryngeal Mask or Single Lumen Endotracheal Tube Before Emergence Following a Thoracic Surgery: a Randomized-controlled Trial.
Brief Title: Benefits of Exchanging a Double Lumen Tube to a Proseal Laryngeal Mask or a Single Lumen Tube After a Thoracic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Issam Tanoubi, Université de Montréal, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Proseal08083
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Cough; Laryngospasm; Apnea; Desaturation; Voice Hoarseness
Keywords: Exchanging double lumen tube with laryngeal mask Proseal; Exchange double lumen tube with tracheal tube; Exchange double lumen tube before emergence decrease cough; thoracoscopy and postoperative respiratory complications; thoracostomy and postoperative respiratory complications; postoperative cough; postoperative respiratory complications; laryngeal mask and postoperative respiratory complications
MeSH Terms: conditions — Cough; Laryngismus; Apnea; Hoarseness | interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): The double lumen tube is kept until extubation; there is no exchange with any tracheal tube or LMA.
- Proseal (Active Comparator): The double lumen tube is exchanged with a Proseal (LMA) before emergence according to the study protocol.
  Interventions: Device: LMA Proseal
- Tracheal tube (Active Comparator): The double lumen tube is exchanged with a tracheal tube before emergence according to the study protocol.
  Interventions: Device: Tracheal tube

INTERVENTIONS:
Device: LMA Proseal — Once surgery is completed, the patient is transferred onto a gurney. Train of four is checked. Patient is ventilated with 100% oxygen. Remifentanil 0.5 ug/ml IV is administered. 30 seconds to 1 minute later, secretions are suctioned. Depth of anesthesia is ensured by deflating, inflating, then deflating the tracheal balloon of the DLT and checking for absence of movement, swallowing, or coughing. The DLT is removed, then the LMA proseal is inserted. Respiratory and hemodynamics parameters are noted. Tolerance of the exchange (presence of cough, movement, laryngospasm, desaturation) is noted. Inhalational gas is stopped. Reversal agent is administered if appropriate. Spontaneous breathing is titrated for <12 with boluses of fentanyl 25ug or sufentanil 2.5ug q 5mins.
  If failure to insert Proseal occurs, a second attempt is made after deepening anesthesia with propofol 1mg/kg and remifentanil 0.5ug/kg IV. If failure occurs again, the patient is intubated with a tracheal tube.
  Other Names: Proseal, laryngeal mask airways
  Arms: Proseal
Device: Tracheal tube — Once surgery is completed, the patient is transferred onto a gurney. Train of four is checked. Patient is ventilated with 100% oxygen. Remifentanil 0.5 ug/ml IV is administered. 30 seconds to 1 minute later, secretions are suctioned. Depth of anesthesia is ensured by deflating, inflating, then deflating the tracheal balloon of the DLT and checking for absence of movement, swallowing, or coughing. The DLT is removed, then a tracheal tube (size 7 for women, size 8 for men) is inserted. Respiratory and hemodynamics parameters are noted. Tolerance of the exchange (presence of cough, movement, laryngospasm, desaturation) is noted. Inhalational gas is stopped. Reversal agent is administered if appropriate. Spontaneous breathing is titrated for <12 with boluses of fentanyl 25ug or sufentanil 2.5ug q 5mins.
  Other Names: Single lumen endotracheal tube
  Arms: Tracheal tube

SUMMARY:
The purpose of this study is to determine whether exchange of the double lumen tube before emergence with a laryngeal mask airway (Proseal) or a tracheal tube will reduce cough at emergence.

DETAILED DESCRIPTION:
Intubation with a double lumen tube is often the preferred method to ensure isolation of the lung and proper exposition of the surgical site during thoracoscopies and thoracostomies. Unfortunately, because of the length and diameter of the double lumen tube, it is known to cause more irritation in the upper airways thereby inducing cough at emergence. In turn, cough has been associated with numerous multisystemic complications. Severe respiratory complications include laryngospasm or upper airway obstruction, desaturation, vocal cord injury, tracheal and bronchial ruptures. The purpose of this study is to determine whether exchange of the double lumen tube before emergence with a laryngeal mask airway (Proseal) or a tracheal tube will reduce cough at emergence.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 year old undergoing elective thoracic surgery
* intubation with double lumen tube required
* patients in category ASA 1, 2, 3

Exclusion Criteria:

* Difficult intubation anticipated
* Presence of gastro-esophageal reflux
* Patients considered with a full stomach
* Body mass index >30
* Presence of nasogastric tube when exchange should be done
* Patients undergoing oesophagogastrectomy
* Allergy to any medication used in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequency of cough | From change to supine position to 10 minutes after removal of airway device

CONTACTS AND LOCATIONS:
Overall Officials: François Donati, PhD MD FRCPC, Study Chair — Université de Montréal; Issam Tanoubi, MD, Study Director — Université de Montréal; Joanna Ng Man Sun, MD, Principal Investigator — Université de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Tanoubi I, Sun JN, Drolet P, Fortier LP, Donati F. Replacing a double-lumen tube with a single-lumen tube or a laryngeal mask airway device to reduce coughing at emergence after thoracic surgery: a randomized controlled single-blind trial. Can J Anaesth. 2015 Sep;62(9):988-95. doi: 10.1007/s12630-015-0403-2. Epub 2015 May 19. PMID 25985845